CLINICAL TRIAL: NCT01907139
Title: Comparative Efficacy Research of Robot-Assisted Therapy With and Without Constraint-Induced Therapy in Stroke Rehabilitation: Does the Combined Therapy Improve Outcomes Compared With Monotherapy?
Brief Title: Comparative Efficacy Research of Robot-Assisted Therapy With and Without Constraint-Induced Therapy in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 01-M07-072
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Cerebrovascular Accident
Keywords: comparative efficacy research; combination therapy; neurorehabilitation; robot-assisted therapy; constraint-induced therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Distributed constraint-induced therapy (dCIT) (Experimental): The dCIT group will focus on restriction on movement of the unaffected hand by placement of the hand in a mitt for 6 hours/day and intensive training of the affected UL in functional tasks for 1.5 hours/weekday over the 4 weeks.
  Interventions: Behavioral: Distributed constraint-induced therapy
- Robot-assisted therapy (RT) (Experimental): The ArmeoSpring (Hocoma AG, Switzerland) will be adopted in this study. It is a 5 degree-of-freedom skeleton mechanism that automates arm movement in a gravity-supported and computer-enhanced environment. The design of the arm support component of the ArmeoSpring is based on Wilmington Robotic Exoskeleton, an antigravity arm support. The ArmeoSpring g provides weight support for the arm across a large 3D workspace, enabling naturalistic movement across approximately 66% of the normal workspace in the vertical plane and 72% in the horizontal plane. Its main structure consists of an arm exoskeleton with elastic bands that relieve the weight of the limb and provide a sense of arm flotation at all positions in the available workspace. A custom grip sensor consisting of a water-filled cylindrical bladder detects grip pressure and finger movement and allows incorporation of grasp and release practice into arm training.
  Interventions: Behavioral: Robot-assisted therapy
- Dose-matched control therapy (DMCT) (Active Comparator): The DMCT group mediated by the therapists will be designed to control for the duration of therapy in amount of therapy hours. This group will received a structured protocol using conventional occupational therapy techniques such as neuro-developmental techniques with emphasis on functional tasks and muscle strengthening.
  Interventions: Behavioral: Dose-matched control therapy
- RT + dCIT (Experimental): In this combination therapy group, the participants will received 2 weeks of RT using the ArmeoSpring and followed by 2 weeks of distributed CIT. The treatment principles of RT and distributed CIT are the same with those described in the monotherapy of RT or dCIT, respectively. This combined intervention group may integrate proximal (shoulder and elbow) to distal (wrist and hand) training of the UL and help transfer from motor ability gained to functional performance improvement. That is, it appears to associate with the advantages/effects of each RT and dCIT intervention.
  Interventions: Behavioral: Robot-assisted therapy; Behavioral: Distributed constraint-induced therapy

INTERVENTIONS:
Behavioral: Robot-assisted therapy — Instrumentation of the ArmeoSpring with position sensors at each joint enables it to be used as a 3D input device for computer game play with the hemiparetic arm. Games were designed to simulate functional arm movements to provide training in a simple virtual reality environment. Vu Therapy games were developed with the goal of enabling repetitive task-specific practice including grocery shopping, cleaning a stovetop, and playing basketball. In this way, stroke patients who are unable to use their severely weakened arms in a functional way are able to practice task-specific movements in a simulated, gravity-reduced environment. Auditory and visual feedback is provided throughout game play to maintain the patient's attention and motivation. In addition, users are provided objective feedback of task performance at the end of each game to enhance motivation and awareness of progress.
  Other Names: RT
  Arms: RT + dCIT; Robot-assisted therapy (RT)
Behavioral: Distributed constraint-induced therapy — The dCIT group will focus on restriction on movement of the unaffected hand by placement of the hand in a mitt for 6 hours/day and intensive training of the affected UL in functional tasks for 1.5 hours/weekday over the 4 weeks. Participants in this group will focus on the intensive training of the affected arm in functional activities with behavioral shaping. The shaping techniques will involve individualized task selection, graded task difficulty (e.g., practicing deficient parts of the selected activity and then performing the entire activity), verbal feedback, prompting, physical assistance with movements, and modeling. The level of challenge will be adapted based on patient ability and improvement. Participants will be also required to place their unaffected hand and wrist in a mitt for 6 hours a day during the 4-week period and document mitt compliance in daily logs.
  Other Names: dCIT
  Arms: Distributed constraint-induced therapy (dCIT); RT + dCIT
Behavioral: Dose-matched control therapy — The DMCT group mediated by the therapists will be designed to control for the duration of therapy in amount of therapy hours. This group will received a structured protocol using conventional occupational therapy techniques such as neuro-developmental techniques with emphasis on functional tasks and muscle strengthening. The treatment protocol will include (1) passive range of motion exercises, stretching of the affected limb, or facilitatory and inhibitory techniques for 15 to 20 minutes, (2) tasks for training fine motor or dexterous function for 20 minutes, (3) arm exercises or gross motor training for 20 minutes, (4) muscle strengthening of the affected UL for 15 to 20 minutes, and (5) activities of daily living or functional tasks practice for 15 to 20 minutes. The activities will be adapted based on the level of motor impairment and individual needs of the patients.
  Other Names: DMCT
  Arms: Dose-matched control therapy (DMCT)

SUMMARY:
There are 3 specific study purposes. First, we will examine the treatment effects of RT combined with dCIT (RT + dCIT) compared to RT, dCIT, and a dose-matched control therapy (DMCT) in stroke patients. Outcome domains will include motor, sensory, and muscle functions, amount of arm activity in real-life situations, patient-reported outcomes of daily performance and quality of life, and kinematic performance. Additionally, potential adverse effects including fatigue, pain, and a biomarker of oxidative stress will be examined. Second, we will investigate if the demographical and clinical characteristics of stroke patients may predict the probability of achieving clinically important changes of treatment outcomes. Thirdly, this study will examine whether the improvements after treatment reach clinically important or not and assess clinimetric properties of the outcome measures.

DETAILED DESCRIPTION:
This research project will investigate the efficacy of RT in sequential combination with dCIT relative to the therapies given alone and study the factors relevant to outcomes prediction to inform clinical practice. There will be 3 primary purposes in this comprehensive research:

Ⅰ. We will examine the effects of RT combined with dCIT (RT + dCIT) compared to RT, dCIT, and a dose-matched control therapy (DMCT) in stroke patients. Outcome domains will include motor, sensory, and muscle functions, amount of arm activity in real-life situations, patient-reported outcomes of daily performance and quality of life, and kinematic performance at before treatment, midterm assessment, and after treatment. In addition, potential adverse effects including post-exertional fatigue, post-exertional pain, and a biomarker of oxidative stress will be examined. We hypothesized that the therapeutic regimen combining RT with dCIT will contribute to more significantly reduction in impairment and disability for stroke patients than the other intervention groups.

Ⅱ. We will investigate if the demographical and clinical characteristics of stroke patients may significantly predict the probability of achieving clinically significant changes of treatment outcomes. The proposed candidate predictors will be chronicity, side of lesion, muscle tone, finger extension, motor function of distal upper limb (UL), and amount of real-life arm activity.

Ⅲ. We will examine whether the improvements after treatments are clinically important and will assess clinimetric properties of the outcome measures to establish the clinical significance relevant for individualized stroke rehabilitation. We will also assess and compare the clinimetric properties (e.g., validity, responsiveness, minimal detectable change, and minimal clinically important difference) of the rehabilitation outcomes to inform selection of instruments.

ELIGIBILITY:
Inclusion Criteria:

* 6 months onset from a first-ever unilateral stroke
* an initial UL subsection of the Fugl-Meyer Assessment score of 20 to 56
* minimal motor criteria to receive CIT (i.e., ≥ 100 wrist extension and ≥ 100 extension at the thumb and any two other digits)
* no excessive spasticity in any of the joints of the affected UL (modified Ashworth scale ≤ 3)
* without upper limb fracture within 3 months
* be able to follow study instructions and perform study tasks (Mini Mental State Examination ≥ 24)
* welling to provide written informed consent

Exclusion Criteria:

* physician-determined major medical problems or poor physical conditions that would interfere with participation
* excessive pain in any joint that might limit participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) | Baseline, 2 weeks, and 4 weeks
  The upper-extremity subscale of the FMA will be used to assess motor impairment. The 33 upper limb items measure the movement and reflexes of the shoulder/elbow/forearm, wrist, hand, and coordination/speed. They are scored on a 3-point ordinal scale (0-cannot perform, 1-performs partially, 2-performs fully). The maximum score is 66, indicating optimal recovery. The sub-score of a proximal shoulder/elbow (FMA s/e: 0-42) and a distal hand/wrist (FMA h/w: 0-24) will be also calculated to investigate the treatment effects on separate upper extremity elements. The reliability, validity, and responsiveness of the FMA in stroke patients have been shown to be good.
Change in Wolf Motor Function Test (WMFT) | Baseline, 2 weeks, and 4 weeks
  The WMFT was originally designed to assess the effects of CIT on the return of arm function for stroke and traumatic brain injury. The assessment requires the participant to perform 15 function-based and 2 strength-based tasks. The tasks are averaged to produce a score in seconds that ranges from 0 to 120 seconds. For functional ability scoring, we used a 6-point ordinal scale where 0 indicates "does not attempt with the involved arm" and 5 indicates "arm does participate; movement appears to be normal." The clinimetrics of the WMFT has been ascertained in stroke patients.
Change in Functional Independence Measure (FIM) | Baseline, 2 weeks, and 4 weeks
  The FIM consists of 18 items grouped into 6 subscales measuring self-care, sphincter control, transfer, locomotion, communication, and social cognition ability. Each item is rated from 1 to 7 (maximum score 126) based on the required level of assistance to perform the tasks (e.g., 1-complete assistance and 7-complete independence). A higher score on any subscale indicates a less disability. The FIM has been shown to have good inter-rater reliability, construct validity, and discriminant validity.
Change in Motor Activity Log (MAL) | Baseline, 2 weeks, and 4 weeks
  The MAL consists of 30 structured questions to interview how the patients rate the frequency (amount of use subscale) and quality (quality of movement subscale) of movements while using their affected arm to accomplish each of the 30 daily activities. The score of each item ranges from 0 to 5, and the higher scores indicate more frequently used or higher quality of movements. The summary score is the mean of the item scores. The clinimetric properties of the MAL in stroke patients have been validated.
Change in Stroke Impact Scale Version 3.0 (SIS 3.0) | Baseline, 2 weeks, and 4 weeks
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. The reliability, validity, and responsiveness have been shown to be satisfactory in stroke patients.

SECONDARY OUTCOMES:
Change in Medical Research Council scale (MRC) | Baseline, 2 weeks, and 4 weeks
  Muscle power of the affected arm will be examined by the MRC scale in this project. The MRC is a commonly used and widely accepted scale. The MRC scale is reliable measurement in stroke patients with score ranged from 0 to 5 Grade of 0 indicates no contraction, 1: flicker or trace contraction, 2: active movement, with gravity eliminated, 3: active movement against gravity, 4: active movement against gravity and resistance, and 5: normal power.
Change in Modified Ashworth Scale (MAS) | Baseline, 2 weeks, and 4 weeks
  The MAS is one of the most frequently used of the clinical scales for assessing muscle spasticity by means of a quick stretch response. Muscle tone of upper limb will be evaluated by the MAS in this project. The scoring of the MAS ranges from 0 (no increase in muscle tone) to 4 (affected part rigid). The inter-rater reliability, intra-rater reliability, and criterion validity of the MAS have been validated in stroke patients.
Change in Revised Nottingham Sensory Assessment (RNSA) | Baseline, 2 weeks, and 4 weeks
  The RNSA includes tactile sensation, kinesthetic sensation, and stereognosis. The RNSA is reliable measure of sensory function in stroke patients. For tactile sensation, the patient will be asked to indicate whenever he or she feels the test sensation. For kinesthetic sensations, all 3 aspects of movement will be tested: appreciation of movement, its direction and accurate joint position sense. The limb on the affected side of the body will be supported and moved by the examiner in various directions but movement is only at one joint at a time. The patients will be asked to mirror the change of movement with the other limb. For stereognosis, the object will be placed in the patient's hand for a maximum of 30 seconds. Identification is by naming, description or by pair-matching with an identical set. The object may be moved around the affected hand by the examiner.
Change in MyotonPRO | Baseline, 2 weeks, and 4 weeks
  The MyotonPRO represents a noninvasive way to characterize the viscoelastic properties of skeletal muscle in vivo. Three measurement parameters in the MyotonPRO: F - Frequency, Hz, characterizes muscle tone; D - Decrement, characterizes muscle elasticity; S - Stiffness, N/m, characterizes muscle stiffness. The working principles of the MyotonPRO are as follows: the testing end of the MyotonPRO will be placed perpendicular to the skin surface above the muscle to be measured, a brief mechanical impulse will be applied, shortly followed by a quick release to the muscle through an acceleration probe, and the damped oscillations of the muscle response will be recorded by the acceleration transducer at the testing end of the device. The oscillation graph creates during the measurement expresses the acceleration of the testing end.
Change in Actigraphy | Baseline, 2 weeks, and 4 weeks
  The activity monitors will be used to provide a direct and objective measure of the amount of the impaired arm movement outside the laboratory. This measure, quantitatively recording the amount of activity in free-living conditions, will be used to reflect increase in the amount of affected arm use over time. The participants will be asked to wear an activity monitor, Actigraphy (Ambulatory Monitoring Inc., New York), on each wrist for 3 consecutive days to measure what amount they actually do in their daily life before and immediately after treatment. The Actigraphy can be attached to the subject's limb and measures the motion of that limb through an accelerometer. In this project, acceleration will be sampled at 10 Hz and summed over a user-specified epoch. The recording epoch will be 2 seconds; recording capacity will be approximately 72 hours. The ratio of affected to non-affected arm movement is a reliable and valid real-life measure of treatment outcome.
Change in Visual analogue scale (VAS) for assessing post-exertional fatigue and pain | From the date of treatment started until the date of treatment ended at 0, 90, 105 minutes for each treatment period
  The visual analogue fatigue scale (VAFS) and visual analogue pain scale (VAPS) will be used to assess the level of post-exertional fatigue and post-exertional pain. The VAS consists of score ranges from 0 to 100 measured in millimeters on a 10-cm vertical line. The scores will be obtained by measuring the lines from "no fatigue" to "very severe fatigue" and from "no pain" to "very severe pain". Post-exertion fatigue will be calculated by subtracting the VAFS at-rest score from the VAFS post-exercise score, and recovery rate was calculated using the formula: (VAFS post-exercise-VAFS post-recovery) / (VAFS post-exercise-VAFS at-rest) ×100). The VAFS has been established to have good reliability, validity, and responsiveness in stroke patients.
Change in Urinary 8-hydroxydeoxyguanosine (8-OHdG) | Baseline, 2 weeks, and 4 weeks
  Urinary 8-OHdG is a stable and integral biomarker of oxidative DNA damage. Urine samples of the patients will be collected before and after intervention, and will be stored at -20 ℃ refrigerator. The urinary 8-OHdG levels will be analyzed with a highly sensitive and selective method, using isotope-dilution liquid chromatography with tandem mass spectrometry (LC/MS/MS), as previously published by Hu et al. (2004). On the basis of previous studies that used the LC/MS/MS analytic method, the mean urinary 8-OHdG levels in the control patients have been reported in the range of 4 to 6 ng/mg creatinine.
Change in Kinematic analysis | Baseline, 2 weeks, and 4 weeks
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University, Taiwan; Yi-shiung Horng, PhD, Principal Investigator — Buddhist Tzu Chi General Hospital Taipei Branch
Locations (1):
- Buddhist Tzu Chi General Hospital Taipei Branch, New Taipei City, Taiwan, Taiwan